CLINICAL TRIAL: NCT06285305
Title: Attitudes and Behaviors of Surgical Intensive Care Nurses Towards End-of-Life Care and Identification of Barriers to End-of-Life Care: A Multicenter Cross-Sectional Study
Brief Title: Surgical ICU Nurses' Attitudes on End-of-Life Care
Status: Not yet recruiting | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Researcher Asisstan, Kilis 7 Aralik University
Other Study IDs: kilis_2
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: PATİENT CARE; Intensive Care Unit
Keywords: End-of-Life Care; Surgical Intensive Care Nurses; Attitudes; Behaviors; Barriers; Intensive Care Unit; Patient Care; Ethical Standards; Quality of Life; Clinical Decision-Making
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to explore the attitudes and behaviors of nurses working in surgical intensive care units (ICUs) towards end-of-life care, alongside identifying the barriers they face in providing such care. Despite the universal need for end-of-life care, with an estimated 56.8 million people requiring it annually, only a fraction receive adequate services. The concept of a "good death" has evolved, now emphasizing patient and family wishes, and aligning with clinical, cultural, and ethical standards. In the U.S., a significant portion of deaths occur in hospitals, often involving surgical interventions in the final stages of life. Nurses in ICUs play a crucial role in delivering end-of-life care, making their attitudes and behaviors pivotal to the quality of care provided. Previous studies have indicated a positive correlation between nurses' attitudes towards end-of-life care and their ethical conduct in care delivery. However, research specifically focusing on surgical ICU nurses and the challenges they encounter in end-of-life care is limited. This study seeks to fill that gap, enhancing understanding of the factors that influence end-of-life care in surgical ICUs and potentially guiding improvements in care practices and policy.

DETAILED DESCRIPTION:
End-of-life care aims to meet the physical, psychological, social, and spiritual needs of patients approaching death and their families, helping people live as well as possible until death, supporting decision-making about the last months of life, and ensuring a dignified death (Filiz 2017). It also encompasses support provided to the family during the illness and care after death to facilitate a healthier grieving process (Karakaya 2020). Every year, an estimated 56.8 million people require end-of-life care, of which 25.7 million are in their last year of life, yet only 14% receive this care (WHO 2020). Everyone has the right to die in peace, just as they have the right to live in peace. The concept of a good death has evolved from being perceived in the past based on different parameters, such as dying at home, dying without pain, dying in a hospital, or dying accompanied by religious rituals (Uğur 2020), to being generally perceived today as a death that is in accordance with the wishes of patients and their families; and is compatible with clinical, cultural, and ethical standards (Granda-Cameron 2012).

In the United States, approximately 2.5 million people die each year, with more than 60% of these deaths occurring in hospitals, and about half of those dying in hospitals do so within three days of admission to an intensive care unit (Cicarello 2003). Surgical intervention is a common practice in the final stages of life, especially among hospitalized patients, with an estimated one-third of patients undergoing surgery in the last month of their life (Taylor 2017). A study conducted by Özkan and Şahinoğlu in 2009 in Turkey found that the one-year mortality rate in the surgical intensive care unit of a university hospital was 46% (Özkan 2009).

Nurses are responsible for the care of patients in the dying process in intensive care units. Therefore, nurses working in intensive care units can encounter death at any moment (Yılmaz 2015). In this context, end-of-life care, which includes the patient and their family, is a natural element of intensive care nursing (Filiz 2017).

An attitude is the storage in the mind of feelings, thoughts, and tendencies towards an object (Yavuz Karamanoğlu 2022). Behavior is the actions and reactions shown by an individual in response to situations (Cengiz 2020). Nurses are influenced by their individual attitudes and behaviors while practicing their profession. The attitudes and personal characteristics of nurses affect their professional competence (Karahan 2018). Therefore, the attitudes and behaviors of nurses towards end-of-life care can affect the quality of life, decision-making processes, and coping skills with death of patients and their families. A study showed that the attitudes and behaviors of intensive care nurses towards end-of-life care are positively related to their ethical attitudes in the care process (Efil 2023). Another study found that nurses' attitudes and behaviors affect their levels of clinical decision-making (Erzincanlı 2021). A strong positive relationship was found between nurses' attitudes and behaviors towards end-of-life care and their personal development, with self-actualized nurses having more positive attitudes and behaviors towards end-of-life care (Cengiz 2020).

Another factor determining the quality and effectiveness of end-of-life care in intensive care is the barriers to end-of-life care. These barriers can be related to the patient or family members, such as communication problems, religious beliefs and cultural differences, emotional and psychological stress experienced by family members. Institutional factors can also affect the effectiveness of end-of-life care, such as restricted family access to intensive care or lack of procedures related to end-of-life care. In addition, clinician-related factors are important, such as inadequate communication skills, unrealistic expectations about prognosis, or stress can affect the quality of end-of-life care (Friedenberg 2011; Xu 2022).

Therefore, identifying the attitudes and behaviors of intensive care nurses towards end-of-life care can be effective in understanding and solving problems that arise in nurses' clinical decision-making processes, the quality of care provided to patients and their families, and ethical issues in end-of-life care practices. Identifying educational and research needs in this area will also be beneficial in developing nurses' decision-making abilities and increasing their levels of dealing with ethical challenges. Additionally, identifying barriers to end-of-life care; can facilitate the reduction of these barriers and the implementation of measures in clinics.

The literature review shows studies examining factors affecting end-of-life care in intensive care, nurses' decision-making processes, ethical issues, and factors related to nurses (Erzincanlı 2021; Cicarello 2003; Yılmaz 2015; Kuşlu 2019; Ranse 2012; Harris 2014; Fridh 2014). However, the number of studies examining the attitudes and behaviors of nurses working in surgical intensive care towards end-of-life care and the barriers to end-of-life care is quite limited. The aim of this study is to examine the attitudes and behaviors of surgical intensive care nurses towards end-of-life care and the barriers to end-of-life care.

ELIGIBILITY:
Inclusion Criteria:

* Nurses working in the Surgical Intensive Care Unit,
* Nurses willing to participate in the study will be included.

Exclusion Criteria:

* Nurses who wish to withdraw from the study at any stage after being included will not have their data included in the research.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population consists of nurses employed in Surgical Intensive Care Units (SICUs) who have voluntarily agreed to participate in this research. This group is targeted due to their direct involvement and experience with end-of-life care practices within a highly specialized and critical care environment. The inclusion of SICU nurses allows for a focused examination of the attitudes, behaviors, and perceived barriers towards end-of-life care in a setting that frequently confronts the complexities of life-threatening conditions and death. This specific population provides valuable insights into the challenges and needs associated with end-of-life care in surgical intensive care contexts, contributing to the development of more effective care strategies and policies to support both patients and healthcare professionals in this sensitive area of medical care.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Descriptive Information Form | up to 20 weeks
  This section contains questions about health professionals' demographic and professional characteristics, such as age, gender, educational background, marital status, and professional experience.
Attitudes and Behaviors Towards End-of-Life Care Scale for Intensive Care Nurses | up to 20 weeks
  Developed by Zomorodi (2008) and revised by Zomorodi and Lynn (2010), this scale measures intensive care nurses' attitudes and behaviors regarding end-of-life care. It has a Cronbach's alpha of 0.78 and was adapted into Turkish by Yalçınkaya (2016) with a reliability of 0.70. The scale, using a five-point Likert type, consists of two sub-dimensions (attitudes and behaviors towards end-of-life care) and includes a total of 16 items.
Barriers to End-of-Life Care in Surgical Intensive Care Form | up to 20 weeks
  Created after reviewing sources (Nelson 2006; Friedenberg 2012; Taylor 2017; Ganz 2019; Diaz 2020; Xu 2022; Gu 2022), this form identifies barriers nurses face in providing end-of-life care in surgical ICUs through 20 structured questions on a five-point Likert scale. The form's content validity was assessed by two intensive care anesthesiologists and three nursing faculty members through email. Items were rated on a scale of 1-4 for appropriateness and clarity (1: not suitable, 2: somewhat suitable, 3: quite suitable but needs minor changes, 4: very suitable). The Content Validity Index (CVI) was calculated as 0.96, indicating the form is suitable for this research (Davis 1993).

CONTACTS AND LOCATIONS:
Locations (1):
- Islam, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Plan to Share IPD:
  Intent: To share de-identified participant data underpinning published results.
  Data Included: De-identified responses to surveys and demographic information.
  Availability: 9 to 36 months post-publication.
  Access: Researchers must submit a proposal evaluated for scientific merit. A data access agreement is required.
  Format: Secure, de-identified, suitable for analysis.
  Documentation: Study protocol, data dictionary, and analysis plan provided.
  Protection: Participant privacy and data confidentiality ensured.
  End of Sharing: Data securely destroyed or archived as per agreement.
  This plan supports open science while protecting participant rights.